CLINICAL TRIAL: NCT00609375
Title: Efficacy of Cefepime Continuous Infusion Versus an Intermittent Dosing Regimen in Adult Critically Ill Patients With Gram Negative Bacilli Bacteremia
Brief Title: Efficacy of Cefepime Continuous Infusion Versus an Intermittent Dosing Regimen
Acronym: CEFPK/PD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Javeriana University (Other)
Collaborators: Asociacion Colombiana de Infectologia, ACIN. Infectious Diseases Society of Colombia (Unknown); Hospital Simon Bolivar, Bogota (Unknown); Clinica Palermo, Bogota (Unknown); Hospital Santa Clara, Bogota (Unknown); Fundación San Carlos, Bogota (Unknown); Hospital san Juan de Dios, Antioquia (Unknown); Hospital san Jorge, Pereira (Unknown)
Responsible Party: Carlos Arturo Alvarez, Medicine School, Pontificia Universidad javeriana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Universidad Javeriana
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2008-02-07 (Estimated); Status verified 2008-01

CONDITIONS: Sepsis; Bacteremia
Keywords: Sepsis; Bacteremia; Intravenous infusions; cefepime
MeSH Terms: conditions — Sepsis; Bacteremia | interventions — Cefepime

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): Administration of cefepime in continuous infusion (3 Gr over 24 hours) for at least 7 days and no more than 14 days days at the discretion of the investigator. Administration of saline solution 0.9%, 50-100 mL over 30 minutes every 8 hours.
  Interventions: Drug: cefepime
- II (Active Comparator): Administration of cefepime in intermittent infusion (1 Gr over 30 minutes every 8 hours) for at least 7 days and no more than 14 days days at the discretion of the investigator.Administration of saline solution 0.9%, 50-250 mL over 24 hours
  Interventions: Drug: cefepime

INTERVENTIONS:
Drug: cefepime — Administration of cefepime in continuous infusion (3 Gr over 24 hours) for 7-14 days at the discretion of the investigator. Administration of saline solution 0.9%, 50-100 mL over 30 minutes every 8 hours.
  Other Names: maxipime
  Arms: I
Drug: cefepime — Administration of cefepime in intermittent infusion (1 Gr over 30 minutes every 8 hours) for 7-14 days at the discretion of the investigator.Administration of saline solution 0.9%, 50-250 mL over 24 hours
  Other Names: Maxipime
  Arms: II

SUMMARY:
To determine the efficacy of the administration of 7 to 14 days of cefepime in a continuous infusion vs an intermittent (every 8 hours) administration, in adult patients hospitalized in Bogotá with sepsis and bacteremia caused by gram negative bacilli. The outcome was the rate of clinical cure and microbiological cure after 7 and 14 days of initiation of therapy and rates of relapse after 28 days.

Hypothesis: The administration of beta lactams in continuous infusion allows a clinical or microbiological cure greater than the intermittent administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sepsis, severe sepsis o septic shock diagnosis hospitalized in Intensive care Unit.
* Presence or suspect of Gram negative bacilli bacteremia
* To be possible the follow up according to planned visits
* Patients should be venous access to administrate the antibiotic
* Patients, whom the physicians consider cefepime like election treatment

Exclusion Criteria:

* Patients with a high degree of immunosuppression defined by:

  * The presence of neutropenia (Neutrophils count less than 500 cells/mL, or Infection with HIV-AIDS with count of less than 50 CD4 cells/mL, or chronic Administration of immunosuppressive drugs (prednisone more than 5 mg/per day, azathioprine, cyclophosphamide, mycophenolate mofetil, etc.)
* Patients with chronic renal failure.
* Pregnant female patients
* Patients in whom to approach the doctor is considered with a high probability of dying in the next 48 hours (e.g. multiorgan system failure with more than 5 organs engaged according to the criteria of MarshalL et al. or shock irreversible.
* Patients with chronic infections as osteomyelitis or have prosthesis that would perpetuate the infection and requiring the administration of antibiotics for an extended time (including Endocarditis). -Patients with mixed infections that include Gram positive microorganisms or fungal infections.
* -Patients who have received in the past 30 days cefepime.
* Patients with presence of a gram negative bacillus resistant to cefepime. -Patients who are not able to identify them a bacillus gram negative.
* Patients who they are not able to confirm the antibiotic susceptibility of gram negative bacillus. -Patients with concomitant with antimicrobial activity for Gram negative bacilli (e.g. fluoroquinolones, aminoglycosides, etc.)
* Patients who have known hypersensitivity to B lactams or cefepime

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To evaluate global mortality rate | 28 days

SECONDARY OUTCOMES:
to evaluate clinical and/or microbiologic relapses | 28 days
To evaluate clinical and bacteriological response | 3 days
to evaluate clinical and bacteriological response | 7 days
to evaluate clinical and bacteriological response | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: carlos A Alvarez, MD, Principal Investigator — Pontificia Universidad Javeriana; Alvaro Ruiz, MD; MSc, Study Chair — Pontificia Universidad Javeriana; Fabian GIL, Msc, Study Chair — Pontificia Universidad Javeriana
Locations (7):
- Colombia (7):
  - Hospital San Juan de Dios, Rionegro, Antioquia
  - Clinica Palermo, Bogotá, DC
  - Fundacion San Carlos, Bogotá, DC
  - Hospital Santa Clara, Bogotá, DC
  - Hospital Simon Bolivar, Bogotá, DC
  - Hospital Universitario san Ignacio, Bogotá, DC
  - Hospital San Jorge, Pareira, Risaralda Department